CLINICAL TRIAL: NCT06229002
Title: Biological, Neuropsychological and Electrophysiological Effect of Transcranial Alternative Current Stimulation at Alpha Frequency (α-tACS) on Stressed Healthy Subjects
Brief Title: Effect of Transcranial Alternative Current Stimulation at Alpha Frequency (α-tACS) on Stressed Healthy Subjects
Acronym: CAF-TAS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2023-A01368-37
Record Dates: First submitted 2023-12-20; First posted 2024-01-29 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2023-12

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo-controlled, randomized parallel arms study including 40 healthy participants who will receive active and placebo α-tACS
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants and experimenters (including α-tACS operator) will not be informed about the nature (active or placebo) of the stimulation they will receive
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active tACS stimulation (Experimental): Transcranial alternative current stimulation (tACS) at alpha frequency Single session of tACS : 30 minutes, 2mA, frequency = 10Hz, both electrodes located on the dorsolateral prefrontal cortex (left and right)
  Interventions: Procedure: Transcranial alternative current stimulation (tACS) at alpha frequency
- Sham stimulation (Placebo Comparator): Single session of tACS sham stimulation : both electrodes located on the dorsolateral prefrontal cortex (left and right) ; real current delivered for the first and last 30s of the total stimulation time (ramp-in and ramp-out)
  Interventions: Procedure: Sham stimulation

INTERVENTIONS:
Procedure: Transcranial alternative current stimulation (tACS) at alpha frequency — Single session of tACS
  Arms: Active tACS stimulation
Procedure: Sham stimulation — Single session of tACS sham stimulation
  Arms: Sham stimulation

SUMMARY:
stress. Notably, several studies reported that stress could alter impulsivity, source monitoring, and time perception.

Several mechanisms are involved in the response to a stress factor, among them the hypothalamic-pituitary-adrenal (HPA) axis. The cortisol reactivity (it means the cortisol secretion after the exposure to a standardized stress factor) is a reliable tool to assess the function of HPA. Cortisol secretion is bidirectionally influenced by the prefrontal cortex (PFC), which is involved in the expression and regulation of stress as well. The asymmetry of the alpha band (AFα) is a well known electrophysiological parameter to assess the function of PFC. More precisely, AFα is arising a growing interest, as it is believed to be correlated with the cortisol reactivity. Modifying this asymmetry could influence the stress response.

Transcranial Alternating Current Stimulation (tACS) consists in delivering a sinusoidal alternating current between two electrodes placed on the scalp at a predefined frequency. Previous studious reported that tACS, if delivered at the alpha frequency, increased the alpha band in the stimulated areas

DETAILED DESCRIPTION:
The study will focus on the effect of tACS at alpha frequency (α-tACS), delivered on the dorsolateral prefrontal cortex, on the response to a stress factor.

In this study, while receiving a single α-tACS session, the participants will complete a standardized stress test combining cognitive stress (mental calculation) and physical stress (cold pressure): the Maastricht Acute Stress Test. The main objective aims at assessing the effect of a single session of tACS at alpha frequency, delivered on the dorsolateral prefrontal cortex, on the cortisol reactivity in healthy stressed subjects. In that study, the influence of α-tACS on other biological ; electrophysiological, neuropsychological parameters relevant for the stress response will be assessed also.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed Men and Women aged between 18 and 45
* If woman, hormonal contraception required
* Having given their written informed consent
* Affiliated with a social security scheme
* French speakers and readers

Exclusion Criteria:

* Contraindication to the exposure to exposure to tACS
* Current psychiatric disorder as classified in the DSM-5
* Regular intake of any psychotropic drug or Beta Blocker
* Recent exposure to a traumatic event
* Any debilitating condition making the experimental procedure not feasible
* Pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-24 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Area under the curve (AUC) of the cortisol secretion after the stress task. | 1 day
  Samples of salivary cortisol will be repeatedly (10 occurences) collected during the experiment. The collection will take place before, during and after the stress task.

SECONDARY OUTCOMES:
Effect of α-tACS on the cortisol awakening response in stressed healthy subjects | 4 days
  Samples of morning salivary cortisol will be collected repeatedly (3 times) before experimental session (including the stress task and the tACS session). A last sample of morning salivary cortisol will be collected the following day
Effect of α-tACS on the molecular reactivity to stress | 1 day
  The expression level of different proteins implicated in the intracellular communication channel after the couple cortisol-glucocorticoid receptor was formed (namely : NR3C1) will be assessed. A blood sample will be collected and the expression level of the relevant genes will be assessed by qPCR
Effect of α-tACS on the molecular reactivity to stress | 1 day
  The expression level of different proteins implicated in the intracellular communication channel after the couple cortisol-glucocorticoid receptor was formed (namely : FKBP4) will be assessed. A blood sample will be collected and the expression level of the relevant genes will be assessed by qPCR
Effect of α-tACS on the molecular reactivity to stress | 1 day
  The expression level of different proteins implicated in the intracellular communication channel after the couple cortisol-glucocorticoid receptor was formed (namely : FKBP5) will be assessed. A blood sample will be collected and the expression level of the relevant genes will be assessed by qPCR
Effect of α-tACS on the molecular reactivity to stress | 1 day
  The expression level of different proteins implicated in the intracellular communication channel after the couple cortisol-glucocorticoid receptor was formed (namely : BAG1) will be assessed. A blood sample will be collected and the expression level of the relevant genes will be assessed by qPCR
Effect of α-tACS on the molecular reactivity to stress | 1 day
  The expression level of different proteins implicated in the intracellular communication channel after the couple cortisol-glucocorticoid receptor was formed (namely : PTGES3) will be assessed. A blood sample will be collected and the expression level of the relevant genes will be assessed by qPCR
Effect of α-tACS on the molecular reactivity to stress | 1 day
  The expression level of different proteins implicated in the intracellular communication channel after the couple cortisol-glucocorticoid receptor was formed (namely : HSP90AA1) will be assessed. A blood sample will be collected and the expression level of the relevant genes will be assessed by qPCR
Effect of α-tACS on the molecular reactivity to stress | 1 day
  The expression level of different proteins implicated in the intracellular communication channel after the couple cortisol-glucocorticoid receptor was formed (namely : HSPA1A) will be assessed. A blood sample will be collected and the expression level of the relevant genes will be assessed by qPCR
Effect of α-tACS on the asymmetry of the alpha band (AFα) in stressed healthy subjects | 1 day
  AFα refers to the average difference in alpha-band activity (typically8-13 Hz) between the left and right frontal areas (F3- F7 versus F4-F8, respectively). For a 5-minute block, AFα will be assessed by EEG recording while the participant is at resting state and only requested to alternatively open and close the eyes, according to a standardized procedure
Effect of α-tACS on the beta band in stressed healthy subjects | 1 day
  The participant will have to complete the Kirby Delay Discounting Task (DDT). Subjects are presented with a series of hypothetical choices of amount of reinforcer to be had instantaneously, and a larger reinforcer available after a fixed delay. (For example : "Would you prefer 37€ today or 80€ in 60 days?" The outcome will be the change in the number of immediate choices between before and after the stress period (ΔDDT) express in percent
Effect of α-tACS on source monitoring in stressed healthy subjects | 1 day
  Source monitoring refers to the cognitive processes involved in making attributions about the origins of mental experiences (for example : was this mental experience dreamt?, imagined?, really perceived? If this was perceived, was it produced by myself or by anybody else?". Two subtypes of source monitoring will be tested : the reality monitoring (RM) and the internal monitoring (IM). In each task the participant will be confronted with a list of words he/she will have to determine the source of. The outcome will be the proportion of false attributions, expressed in percent
Effect of α-tACS on impulsivity in stressed healthy subjects | 1 day
  The participant will have to complete the Kirby Delay Discounting Task (DDT). Subjects are presented with a series of hypothetical choices of amount of reinforcer to be had instantaneously, and a larger reinforcer available after a fixed delay. (For example : "Would you prefer 37€ today or 80€ in 60 days?") The outcome will be the change in the number of immediate choices between before and after the stress period (ΔDDT) express in percent
Effect of α-tACS on time perception in stressed healthy subjects | 1 day
  time perception refers to how the brain represents the temporal structure of events and of our environment. This ability can be assessed through different experimental designs. In this protocol, the participants will complete a time reproduction task, consisting in tapping at a defined frequency (1Hz) with a push-button. After a training phase (pressing the push-button while being guided), the participant will have to produce the same rhythm on his own. The outcome will be the mean difference between the reference interval (1s) and the time intervals executed by the participant, express in milliseconds

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Le Vinatier, Bron, AURA, France

IPD SHARING:
Plan to Share IPD: Undecided